CLINICAL TRIAL: NCT01521728
Title: Trial of Resistance and Endurance Exercise in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Nicholas Maragakis, MD, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NA_00022650
Record Dates: First submitted 2012-01-24; First posted 2012-01-31 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Exercise; Resistance; Endurance
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Activity | interventions — Resistance Training; Range of Motion, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Resistance Exercise (Active Comparator): Resistance will be administered using a series of adjustable cuff weights for the upper limbs and hip flexion. Knee flexion and extension will be administered with a weight bench using a leg exercise attachment and free weights.
  Interventions: Other: Resistance Exercise
- Endurance Exercise (Active Comparator): Endurance will be administered using a minicycle. It can be used from a sitting position (chair or wheelchair) for lower limb exercise and then placed on a tabletop for upper limb use.
  Interventions: Other: Endurance Exercise
- Stretching/Range-of-Motion Exercise (Active Comparator): In ALS, stretching and range of motion are routinely recommended for the prevention of "frozen shoulder syndrome" and contractures resulting from weakness. The problem is compounded in ALS where upper motor neuron dysfunction may result in spasticity and incapacitating contractures with pain. Therefore, maintaining an aggressive program for stretching and range of motion exercise is widely accepted as a "standard of care" for ALS management.
  Interventions: Other: Stretching/Range-of-Motion

INTERVENTIONS:
Other: Resistance Exercise — Resistance will be administered using a series of adjustable cuff weights for the upper limbs and hip flexion. Knee flexion and extension will be administered with a weight bench using a leg exercise attachment and free weights.
  Arms: Resistance Exercise
Other: Endurance Exercise — Endurance will be administered using a minicycle. It can be used from a sitting position (chair or wheelchair) for lower limb exercise and then placed on a tabletop for upper limb use.
  Arms: Endurance Exercise
Other: Stretching/Range-of-Motion — Stretching and range of motion exercise is widely accepted as a "standard of care" for ALS management.
  Arms: Stretching/Range-of-Motion Exercise

SUMMARY:
The first questions asked by patients with a new diagnosis of Amyotrophic Lateral Sclerosis (ALS) often include: "Does exercise help slow the progression of the disease?", "Is there any harm in exercising?", or "What type of exercise (endurance or resistance) is most appropriate?" At this time, however, there is a lack of answers for people who suffer from an illness that affects their strength above all else. Yet the beneficial effects of exercise in both healthy people as well as people with other diseases have been extensively studied and resulted in recommendations about the types of exercise that are beneficial. In this study the investigators will ask participants with ALS to exercise in one of three ways: weightlifting (resistance exercise), stationary bicycling (endurance exercise), and range of motion exercise (the current "standard of care" for ALS patients). The investigators will use several different types of tests to determine whether one type of exercise is tolerated better and is safer than another. The investigators will also collect information about how the body responds to exercise in ALS. This study will help in the development of a larger national study to understand how exercise can be combined with other treatments to potentially improve strength and alter the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with familial or sporadic ALS diagnosed as possible, laboratory-supported probable, probable, or definite according to the WFN El Escorial criteria
2. Participants who are ages 18-80, inclusive.
3. Slow Vital Capacity (SVC) must be equal to or greater than 70% of predicted value
4. ALSFRS-R score >30.
5. Patients who are currently on any medications must be on a stable dose for the past 30 days.
6. Participants must provide informed consent prior to completion of any study procedures.

Exclusion Criteria:

1. Participants who are already performing >30 min. of endurance exercise/day for ≥ 3x/week (Borg scale-- "hard" or "somewhat hard") within 30 days of screening.
2. Participants who are already performing resistance exercise ≥ 3x/week within 30 days of screening.
3. Neurologic

   * Participants with history of ALS symptoms over 5 years duration
   * Inability to obtain consent (psychiatric or dementing illness)
   * History of neuromuscular dysfunction not related to ALS
4. Cardiac

   * Patents with clinically significant ECG abnormalities
   * Uncontrolled hypertension (SBP>160 or DBP>110)
   * Recent history of angina (within the last 2 years)
   * Recent history of abnormal stress test (within the last 2 years)
   * Symptomatic severe aortic stenosis
   * Active endocarditis
   * Symptomatic heart failure
5. Respiratory

   * Subjects with a history of respiratory dysfunction not related to ALS (i.e. COPD)
6. General

   * Subjects with chronic infectious disease including HIV, hepatitis B or C.
   * History of substance abuse within the past year
   * Patients who have a history of poor compliance to medical regimens or study requirements.
   * Uncontrolled diabetes
   * Recent embolism (within the last 6 months)
   * Severe orthopedic conditions that would prohibit exercise
7. Pregnancy

   * Female subjects who are pregnant or planning to become pregnant.
   * Female subjects of childbearing potential who are not practicing contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Resistance Exercise Tolerability | 6 months
  Evaluate the tolerability of RESISTANCE exercise in ALS subjects as measured by their ability to complete a 6 month study of a resistance exercise regimen.
Endurance Exercise Tolerability | 6 months
  Evaluate the tolerability of ENDURANCE exercise in ALS subjects as measured by their ability to complete a 6 month study of an endurance exercise regimen.

SECONDARY OUTCOMES:
Vital Capacity | 6 months
  Evaluate the effect of resistance and endurance exercise on slow vital capacity (SVC)
ALS Functional Rating Scores | 6 months
  Evaluate the effect of resistance and endurance exercise on patients scores of the ALS Functional rating scale-revised (ALSFRS-R)
Muscle Strength | 6 months
  Evaluate the effect of resistance and endurance exercise on measures of muscle strength
Spasticity | 6 months
  Evaluate the effect of resistance and endurance exercise on spasticity
Fatigue | 6 months
  Evaluate the effect of resistance and endurance exercise on fatigue
Quality of Life | 6 months
  Evaluate the effect of resistance and endurance exercise on patient quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas M Maragakis, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - Carolinas Medical Center, Charlotte, North Carolina